CLINICAL TRIAL: NCT03842761
Title: Randomized, Double-blind, Placebo-controlled Trial to Investigate Safety, Tolerability, and Pharmacokinetics of Multiple Rising Oral Doses of BI 685509 Over 28 Days in Patients With Mild and Moderate Hepatic Impairment and of Single Oral BI 685509 Dose Compared to Healthy Volunteers
Brief Title: A Study to Test How Different Doses of BI 685509 Are Tolerated in Patients With Liver Problems
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1366-0020
Record Dates: First submitted 2019-02-13; First posted 2019-02-15 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Healthy; Hepatic Insufficiency
MeSH Terms: conditions — Hepatic Insufficiency

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose group 1 (Experimental): Low Dose
  Interventions: Drug: BI 685509; Drug: Placebo
- Dose group 2 (Experimental): Medium Dose
  Interventions: Drug: BI 685509; Drug: Placebo
- Dose group 3 (Experimental): High Dose
  Interventions: Drug: BI 685509; Drug: Placebo
- Dose Group 4 (Experimental): Dose for healthy volunteers dependent on results from prior dose groups with patients
  Interventions: Drug: BI 685509; Drug: Placebo

INTERVENTIONS:
Drug: BI 685509 — Tablet
Drug: Placebo — Tablet

SUMMARY:
The primary objective of this trial is the evaluation of safety and tolerability in patients with mild to moderate hepatic impairment [Child-Turcotte-Pugh (CTP) classification A and B] over different dose regimes of BI 685509 compared to placebo. A secondary objective is to investigate pharmacokinetics of different doses of BI 685509 in patients with mild to moderate hepatic impairment (CTP A and CTP B). In addition, another secondary objective is to compare safety, tolerability, and pharmacokinetics in patients with mild to moderate hepatic impairment (CTP A and CTP B) of single BI 685509 dose to individually matched healthy volunteers

ELIGIBILITY:
Key Inclusion Criteria for all trial participants:

* Age ≥ 18 years at Screening
* Male or female. Women of childbearing potential (WOCBP) participants and male participants able to father a child must be ready and able to use a highly effective method of birth control per ICH M3 (R2) that results in a low failure rate of less than 1% per year when used consistently and correctly throughout the Trial
* Mean Arterial Pressure (MAP) ≥ 85 mmHg at screening visit
* Estimated Glomerular Filtration rate (eGFR) > 70 mL/min/1.73m² according to the CKD-EPI formula at screening visit
* Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial

Key inclusion for Patient Groups 1 and 2

* If on treatment with non-selective beta blockers (NSBB), stable dose since ≥ 8 weeks prior to screening, with no planned dose change of the therapy during study conduct. All other medications stable 4 weeks prior to screening.
* Patient Group 1: Patients with CTP A and portal hypertension (defined as liver stiffness >15 kPa during screening) and without a previous decompensation event [ascites, variceal hemorrhage, encephalopathy, or jaundice (except Gilbert's disease or hemolysis when bilirubin will be almost exclusively indirect hyperbilirubinemia)]. Self-limited and resolved historical events of decompensation like ascites or encephalopathy are allowed if they have occurred at least 6 weeks prior to screening and do not require continued therapeutic intervention at the time of screening.
* Patient Group 2: Patients with CTP B (with liver stiffness >15 kPa during screening)

Key inclusion for Healthy Volunteer group

* Subjects who are healthy, according to the investigator's assessment, individually matched to a participant among Patient Groups 1 and 2 according to the following criteria: age within ± 5 years, body weight within ± 15%, and gender
* Further inclusion criteria apply

Key exclusion for all trial participants

* Ongoing chronic alcohol or drug use, which in the investigator's opinion, makes the patient an unreliable trial participant or unlikely to complete the trial.
* History of relevant orthostatic hypotension, fainting spells, or blackouts based on the investigator´s judgment

Key exclusion for Patient Groups

* Patient Group 2: treatment-refractory ascites
* Patient Group 2: recent decompensation event (refractory ascites, recurrent variceal hemorrhage, recurrent hepatic encephalopathy, spontaneous bacterial peritonitis or hepatorenal syndrome) within 6 weeks of screening
* Further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2021-05-20 (Actual)

PRIMARY OUTCOMES:
The percentage of subjects with drug-related Adverse Events (AEs) among different dose regimes over each up-titration | Up to day 28

SECONDARY OUTCOMES:
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to time of the last quantifiable data point) | Baseline and Up to 72 hours
Cmax (maximum measured concentration of the analyte in plasma) | Up to 72 hours
AUCτ,ss (area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ) [AUCτ,ss will be AUC0-12,ss for bid dosing] | Up to 72 hours
Cmax,ss (maximum measured concentration of the analyte in plasma at steady) | Up to 72 hours
Change from baseline in seated systolic blood pressure (SBP) | Baseline and Up to 28 days
Change from baseline in seated diastolic blood pressure (DBP) | Baseline and Up to 28 days
Change from baseline in heart rate (HR) | Baseline and Up to 28 days
Change from baseline in body weight | Baseline and Up to 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- American Research Corporation at the Texas Liver Institute, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com